CLINICAL TRIAL: NCT01198262
Title: GeneXpert in Studying Staphylococcus Aureus Infections at the Michael E. DeBakey Medical Center, Houston, Texas
Brief Title: Rapid Test to Detect Staphylococcus Aureus in Blood and Wound Infections
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other); Cepheid (Industry)
Responsible Party: Daniel M Musher, Michael E. DeBakey VA Medical Center
Other Study IDs: H-23059
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2008-10

CONDITIONS: Staphylococcus Aureus; Staphylococcal Skin Infections; Bacteremia
Keywords: polymerase chain reaction
MeSH Terms: conditions — Staphylococcal Infections; Staphylococcal Skin Infections; Bacteremia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the Cepheid GeneXpert system accurately detects Methicillin-Resistant and -Susceptible Staphylococcus aureus in blood cultures and wound swabs.

DETAILED DESCRIPTION:
Staphylococcus aureus (SA) remains a major pathogen for human beings, causing infections of skin, soft tissue, bone, and other organs. Bacteremia due to this organism is common, and often occurs in association with medical interventions such as intravenous lines and implantable devices. With the increase in methicillin-resistant S. aureus (MRSA), there has been increasing dependence upon vancomycin, a drug that is inferior to the beta-lactams in its activity against methicillin-susceptible S. aureus (MSSA). If the microbiology laboratory had the ability to identify S. aureus (SA) and its drug susceptibility within hours rather than days, focused therapy would be possible earlier in the course of illness. Clinicians would be able to discontinue antibiotics when SA is not present, to discontinue other broad-spectrum antibiotics when SA is present, or to replace empiric vancomycin with nafcillin when MSSA is identified.

The GeneXpert system (Cepheid) uses real-time PCR to detect genes that encode Staphylococcus aureus protein A (SPA), the staphylococcal cassette chromosome (SCC) and methicillin resistance (mecA). All blood cultures with Gram stain revealing Gram positive cocci in clusters will be tested by PCR the day they became positive. Wound swabs submitted for routine bacteriologic culture will be tested within 48 hr of collection. Results will be compared with those of standard bacteriologic culture. In addition, discrepancies between the GeneXpert and wound culture results will be reviewed in the medical record to ascertain whether antibiotic use at the time of specimen collection is associated with false positive results in which the wound culture yields no S. aureus but PCR detects staphylococcal DNA components.

In the second phase of the study, PCR results for wound swabs and blood cultures will be reported to physicians immediately upon completion of the reaction. The clinical impact of early identification of S. aureus will be determined by comparing antibiotic treatment and clinical outcome of patients for whom early identification was available with those of patients for whom conventional bacteriological culture was the sole diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* Positive blood culture with Gram stain revealing Gram positive cocci in clusters
* All wound swabs submitted to the microbiology lab for standard bacteriologic culture may be included.

Exclusion Criteria:

* Blood cultures that became positive more than 24 hours previously
* Wound swabs for which over 48 hours have passed from the time of collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult and geriatric patients at the Michael E. DeBakey VA Medical Center for have suspected blood and wound infections.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
concordance between PCR results and those of standard bacteriologic culture | 1 year

SECONDARY OUTCOMES:
Impact of early identification of S. aureus on the antibiotics prescribed by physicians and subsequent clinical outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, MD, Principal Investigator — Michael E. DeBakey VA Medical Center; Mark Parta, MD, Study Chair — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States